CLINICAL TRIAL: NCT05757609
Title: Innovative Non-invasive Brain Stimulation in the Rehabilitation of Patients With Chronic Low Back Pain
Brief Title: Transcranial Stimulation for Physiotherapy Optimisation - Chronic Low Back Pain (STOP-CLBP)
Acronym: STOP-CLBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephane ARMAND (Other)
Collaborators: La Tour Hospital (Other); School of Health Sciences Geneva (Other)
Responsible Party: Sponsor-Investigator, Stephane ARMAND, professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-D0077
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Chronic Low Back Pain
Keywords: tDCS; Physiotherapy; Flexion relaxation Phenomenon; prefrontal cortex
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statiticians will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS combined with active physiotherapy (Experimental): transcranial Direct Current Stimulation (tDCS) will be applied for 20 min at an intensity of 2 mA with anodal stimulation targeting the left dorsolateral prefrontal cortex (DLPFC).
  This will be done during a cycling session and will be followed by a physiotherapy program including strengthening and mobilisation exercises.
  It will be applied 3 times a week during 3 weeks.
  Interventions: Device: Anodal tDCS combined with active physiotherapy
- Sham tDCS combined with active physiotherapy (Sham Comparator): Sham transcranial Direct Current Stimulation (tDCS) will be applied for 20 min and this induces similar sensations for the patients, but no change in excitability.
  This will be done during a cycling session and will be followed by a physiotherapy programme including strengthening and mobilisation exercises.
  It will be applied 3 times a week during 3 weeks.
  Interventions: Device: Sham anodal tDCS combined with active physiotherapy

INTERVENTIONS:
Device: Anodal tDCS combined with active physiotherapy — anodal tDCS over prefrontal cortex combined with active physiotherapy
  Other Names: transcranial Direct Current Stimulation; Soterix Medical mini-CT
  Arms: tDCS combined with active physiotherapy
Device: Sham anodal tDCS combined with active physiotherapy — Sham anodal tDCS over prefrontal cortex combined with active physiotherapy
  Other Names: Soterix Medical mini-CT
  Arms: Sham tDCS combined with active physiotherapy

SUMMARY:
The main objective of this study is to investigate the effects of non-invasive brain stimulation (the so-called transcranial direct current stimulation ; tDCS) combined with an active physiotherapy program on the multidimensional impact of pain in patients with Chronic Low Back Pain (CLBP).

The secondary objectives are to compare the effects of these interventions on fear of movement, psycho-emotional state, function, functional connectivity of the left dorsolaterla prefrontal cortex (DLPFC) and erector spinae activity.

Participants will perform:

* 2 sessions including clinical assessments including questionnaires, brain activity assessment (with EEG), and back muscle activity assessment (with EMG)
* 9 interventional sessions of active physiotherapy combined with active or sham tDCS during 3 weeks (3 per week).

Investigators will compare active tDCS with sham tDCS (non active) to evaluate if active tDCS is more effective than sham tDCS.

DETAILED DESCRIPTION:
Previous studies showed that transcranial Direct Current Stimulation (tDCS) targeting specific brain areas may offer novel treatment options in patients with chronic pain, in particular in chronic lower back pain (CLBP). Numerous tDCS trials have shown no evidence of moderate or severe adverse effects, highlighting tDCS as a safe, adequate tolerability and acceptability medical device.

However, several major limits remain before the investigators can start to design larger scale trials and more widespread clinical applications: the lack of knowledge on which brain region to target and about how neural activity is influenced by tDCS in this specific patient's population.

In consequence, the investigators do not know which setup of tDCS they can propose to CLBP patients. For instance, if the investigators manipulate brain interactions at the "wrong" tDCS setting, this may result in limited or no improvement of clinical deficits. Most existing randomized controlled trials (RCT) on tDCS treatment indeed show highly mixed effects which are likely due to incomplete understanding of tDCS-induced changes in brain and behavior. In addition, the majority of RCT have applied tDCS over the primary motor cortex (M1). Furthermore, the targeting of this brain region has recently been questioned and the dorsolateral prefrontal cortex (DLPFC) have been suggested as a valuable alternative. Knowing the mechanisms of action of tDCS based on the new rationale (i.e., tDCS targeting DLPFC) would allow us to define setup which are more likely to succeed.

The primary objective of this study is to investigate the effects of repeated sessions of tDCS combined with active physiotherapy on the multidimensional impact of pain at the end of the intervention compared to sham tDCS with active physiotherapy.

The secondary objectives are to compare the effects of these interventions on fear of movement, psycho-emotional state, function, functional connectivity of the left dorsolateral prefrontal cortex (DLPFC) and erector spinae activity.

The investigators hypothesise that tDCS combined with active physiotherapy will have a greater effect at the end of the intervention and at 3 and 6 months follow-up on all outcomes compared to sham tDCS combined with active physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent,
* ability to follow protocol instructions,
* diagnosis of Non Specific Chronic Low Back Pain ≥12 weeks,
* low back pain with or without radiation to the knee,
* average pain of the previous week ≥ 3 on the VAS (Visual Analogue Scale).
* have sufficient cognitive ability to fill in the various questionnaires (Level B2 French),

Exclusion Criteria:

* herniectomy within the last 6 months,
* lumbar spinal surgery with material (e.g. prosthesis, spondylodesis),
* sensory or motor deficit of a lower limb,
* radiant pain in the lower limb beyond the knee,
* neuropathic pain (according to the dn4 questionnaire),
* diagnosis of an inflammatory rheumatic disease (e.g. rheumatoid arthritis, spondyloarthropathy),
* diagnosis of a chronic generalized pain syndromee of fibromyalgia,
* pregnancy,
* presence of neurological or neuropsychiatric disorders,
* have epilepsy or a recent or severe head injury,
* metal implant in the skull (excluding fillings),
* presence of a pacemaker,
* unhealed wound or skin disease on the skull (electrode contact area)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Core Outcome Measures Index (COMI) | Change from baseline (T0) to immediately after the treatment period (T1)
  The Core Outcome Measures Index (COMI) comprises a short set of questions used to assess the impact of spinal disorders on multiple patient-orientated outcome domains. It is based on a set of individual items selected from established questionnaires and recommended for standardized use by an international group of experts in the field. It consists of seven items to assess the extent of the patient's back pain and leg pain, difficulties with functioning in everyday life, symptom-specific well-being, general quality of life, and social and work disability. A summary index score from 0 (best health status) to 10 (worst health status) can be computed by averaging the values of the five subscales.
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome.

SECONDARY OUTCOMES:
Core Outcome Measures Index (COMI) | Change from baseline (T0) to three months (T2) and six months after the inclusion (T3)
  The Core Outcome Measures Index (COMI) comprises a short set of questions used to assess the impact of spinal disorders on multiple patient-orientated outcome domains. It is based on a set of individual items selected from established questionnaires and recommended for standardized use by an international group of experts in the field. It consists of seven items to assess the extent of the patient's back pain and leg pain, difficulties with functioning in everyday life, symptom-specific well-being, general quality of life, and social and work disability. A summary index score from 0 (best health status) to 10 (worst health status) can be computed by averaging the values of the five subscales.
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome.
Numerical Pain Rating Scale | Change from baseline (T0) to immediately after the treatment period (T1) and three months (T2) and six months after the inclusion (T3)
  Numerical Pain Rating Scale assesses the level of pain on a range from 0 to 10, with 0 being no pain and 10 being the maximum possible pain. For a clinically relevant difference to exist, there has to be a difference between measurements of at least 2 points.
  This scale has been shown to have good levels of reliability for pain measurement.
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome.
Change from Oswestry Disability Index (ODI) | Change from baseline (T0) to immediately after the treatment period (T1) and three months (T2) and six months after the inclusion (T3)
  Oswestry Disability Index (ODI) will be used to analyze the quality of life in people with low back pain. This instrument contains in 10 items that assess the impact of low back pain on several functional activities. Values range from 0 to 5, the highest value indicating greater disability. The end result is the sum of all items.
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome.
Fear Avoidance Beliefs Questionnaire (FABQ) | Change from baseline (T0) to immediately after the treatment period (T1) and three months (T2) and six months after the inclusion (T3)
  Consists of 16 items a self-report questionnaire based on evaluation on the Fear-avoidance model.The maximum score is 96, that representing higher levels of fear-avoidance beliefs. The FABQ has two subscales: the work subscale (FABQw),and the physical activity subscale (FABQpa).
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome
Pain Catastrophizing as assessed by the Pain Catastrophizing Scale | Change from baseline (T0) to immediately after the treatment period (T1) and three months (T2) and six months after the inclusion (T3)
  The Pain Catastrophizing Scale (PCS) is a 13 item survey assessing catastrophizing in context to pain. There are 13 items with 5-pt Likert responses.
  There are several subscales. Scoring Procedure: The PCS total score is computed by summing responses to all 13 items (0-52).
  Subscales:
  Rumination: Sum of items 8, 9, 10, 11 (0-16). Magnification: Sum of items 6, 7, 13 (0-12). Helplessness: Sum of items 1, 2, 3, 4, 5, 12 (0-24).
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome.
Hospital Anxiety Depression Scale (HADS) | Change from baseline (T0) to immediately after the treatment period (T1) and three months (T2) and six months after the inclusion (T3)
  A questionnaire which has also been validated and translated into French. This scale has 14 items, 7 for anxiety subscale and 7 for depression. For each item there is a score of 0 to 3, with a total of 21 points for the scale.
  Scoring is done by completing one trial.
  Continuous measure, lower values indicate better outcome.
Flexion Relaxation Ratio (FRR) on erector spinae | Change from baseline (T0) to immediately after the treatment period (T1)
  Flexion-relaxation ratio is calculated by dividing muscle activity (sEMG) during trunk flexion by muscle activity during full-flexed position. sEMG of lumbar paraspinal muscles is recorder through surface electromyogramm (sEMG) during every trials of each session.
  Scoring is done by completing three trials and calculating the average of the three trials to calculate the Flexion Relaxation Ratio (FRR).
Functional connectivity from Electroencephalogram (EEG) recordings | Change from baseline (T0) to immediately after the treatment period (T1)
  Resting state Electroencephalogram (EEG) functional connectivity (FC) analysis will be calculated.The absolute imaginary component of coherence between Dorso Lateral Prefrontal Cortex (DLPFC) (left and right) and the rest of the brain will be subsequently calculated as index of functional connectivity.
  Continuous measure, higher values indicate better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Armand, Pr, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitals Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knotkova H, Hamani C, Sivanesan E, Le Beuffe MFE, Moon JY, Cohen SP, Huntoon MA. Neuromodulation for chronic pain. Lancet. 2021 May 29;397(10289):2111-2124. doi: 10.1016/S0140-6736(21)00794-7. PMID 34062145
- [Background] Wen YR, Shi J, Hu ZY, Lin YY, Lin YT, Jiang X, Wang R, Wang XQ, Wang YL. Is transcranial direct current stimulation beneficial for treating pain, depression, and anxiety symptoms in patients with chronic pain? A systematic review and meta-analysis. Front Mol Neurosci. 2022 Dec 1;15:1056966. doi: 10.3389/fnmol.2022.1056966. eCollection 2022. PMID 36533133
- [Background] Pinto CB, Teixeira Costa B, Duarte D, Fregni F. Transcranial Direct Current Stimulation as a Therapeutic Tool for Chronic Pain. J ECT. 2018 Sep;34(3):e36-e50. doi: 10.1097/YCT.0000000000000518. PMID 29952860
- [Background] Alwardat M, Pisani A, Etoom M, Carpenedo R, Chine E, Dauri M, Leonardis F, Natoli S. Is transcranial direct current stimulation (tDCS) effective for chronic low back pain? A systematic review and meta-analysis. J Neural Transm (Vienna). 2020 Sep;127(9):1257-1270. doi: 10.1007/s00702-020-02223-w. Epub 2020 Jul 9. PMID 32647923
- [Background] Kandic M, Moliadze V, Andoh J, Flor H, Nees F. Brain Circuits Involved in the Development of Chronic Musculoskeletal Pain: Evidence From Non-invasive Brain Stimulation. Front Neurol. 2021 Aug 31;12:732034. doi: 10.3389/fneur.2021.732034. eCollection 2021. PMID 34531819
- [Background] Luedtke K, May A, Jurgens TP. No effect of a single session of transcranial direct current stimulation on experimentally induced pain in patients with chronic low back pain--an exploratory study. PLoS One. 2012;7(11):e48857. doi: 10.1371/journal.pone.0048857. Epub 2012 Nov 26. PMID 23189136
- [Background] O'Connell NE, Cossar J, Marston L, Wand BM, Bunce D, De Souza LH, Maskill DW, Sharp A, Moseley GL. Transcranial direct current stimulation of the motor cortex in the treatment of chronic nonspecific low back pain: a randomized, double-blind exploratory study. Clin J Pain. 2013 Jan;29(1):26-34. doi: 10.1097/AJP.0b013e318247ec09. PMID 23221623
- [Background] Hazime FA, de Freitas DG, Monteiro RL, Maretto RL, Carvalho NA, Hasue RH, Joao SM. Analgesic efficacy of cerebral and peripheral electrical stimulation in chronic nonspecific low back pain: a randomized, double-blind, factorial clinical trial. BMC Musculoskelet Disord. 2015 Jan 31;16(1):7. doi: 10.1186/s12891-015-0461-1. PMID 25636503
- [Background] Straudi S, Buja S, Baroni A, Pavarelli C, Pranovi G, Fregni F, Basaglia N. The effects of transcranial direct current stimulation (tDCS) combined with group exercise treatment in subjects with chronic low back pain: a pilot randomized control trial. Clin Rehabil. 2018 Oct;32(10):1348-1356. doi: 10.1177/0269215518777881. Epub 2018 May 21. PMID 29783893
- [Background] Pacheco-Barrios K, Cardenas-Rojas A, Thibaut A, Costa B, Ferreira I, Caumo W, Fregni F. Methods and strategies of tDCS for the treatment of pain: current status and future directions. Expert Rev Med Devices. 2020 Sep;17(9):879-898. doi: 10.1080/17434440.2020.1816168. Epub 2020 Sep 15. PMID 32845195